CLINICAL TRIAL: NCT02754622
Title: A Pilot Observational Cohort Study Examining the Feasibility of Measuring Energy Expenditure During Physical Rehabilitation In Critically Ill Patients
Brief Title: The Feasibility of Measuring Energy Expenditure During Physical Rehabilitation In Critically Ill Patients
Acronym: ENERGY-ICU
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/LO/0076
Record Dates: First submitted 2016-04-07; First posted 2016-04-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Intensive Care
Keywords: Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Group: * 2hours before planned physical rehabilitation patients will have their regular ventilator changed to the study ventilator by an ICU Consultant and patients will be clinical stable for 30mins prior to the start of the planned physical rehabilitation.
  * Intended physical rehabilitation as planned will continue without change. This session will be observed by a member of the research team to ensure accurate documentation of the exact timing of performance of the physical rehabilitation activity.
  * Patients will also undergo an assessment by the Medical Research Council Sum-score and maximal inspiratory pressure (all part of routine physiotherapy assessment).
  * Following the physical rehabilitation session, the patient to rate their perceived exertion then patients will also undergo ultrasound assessment of peripheral skeletal muscle architecture.
  * Patients return to their original ventilator after 30mins by an ICU Consultant.
  Interventions: Other: Observational Group

INTERVENTIONS:
Other: Observational Group — Indirect calorimetry measurement during Physical Rehabilitation. Observing planned physical rehabilitation session to determine the rehabilitation activity achieved with IC utilised to determine the number of calories used per session

SUMMARY:
Many patients who are admitted to the intensive care unit (ICU) experience muscle weakness. This muscle weakness occurs whilst patients are unconscious, immobile in bed and on a breathing machine (ventilator). It can develop very quickly, as soon as they become unwell. The investigators know that this weakness can make it harder for patients to regain their normal level of functional ability, such as standing and walking independently. Physical rehabilitation, delivered by physiotherapists, is important for patients as they recover from their critical illness to help them regain strength and to practice the ability to perform physical activities. These activities include sitting on the edge of the bed, standing, stepping on the spot and walking.

However it is difficult to know how hard it is for patients who are recovering from critical illness to perform these types of activities - in other words, how much energy is required. Some patients may find certain activities harder or easier than others. By knowing the energy requirements of patients whilst they take part in different physical rehabilitation activities, physiotherapists may be able to be more accurate with prescribing exercises and designing rehabilitation sessions for patients to practice achieving those activities.

In this study, the investigators will measure the energy requirements of the patients when they take part in physiotherapy-led physical rehabilitation they will have during their admission. To do this, the investigators will use a different ventilator to the one normally used to help their breathing. This ventilator works in exactly the same way, but has an extra component built into it to measure energy requirements. After the rehabilitation session, the patient will return to using their normal ventilator.

DETAILED DESCRIPTION:
Admission to the intensive care unit (ICU) with critical illness is typically associated with profound physical impairments including peripheral skeletal muscle wasting and dysfunction. These effects demonstrate a rapid onset from the point of ICU admission, affect those with higher illness acuity to greater levels, and contribute to the development of intensive care unit-acquired weakness (ICU-AW) defined as severe upper and lower limb muscle weakness. Clinically patients present with significant limitations in exercise capacity and performance of physical functional activities, with deficits persisting for many years following resolution of the original illness.

Physical rehabilitation is recommended to address the physical and functional deficits associated with ICU-AW, and delivery is advocated across the continuum of the patient recovery pathway, commencing whilst in the ICU, following transfer to the ward and beyond hospital discharge. Physical rehabilitation within the ICU typically incorporates early mobilisation (EM), characterised by a hierarchical progression of increasingly functional activities such as active-assisted bed exercises, sitting-on-the-edge-of-the-bed (SOEOB), standing, marching-on-the-spot and walking. These activities are summarised in the ICU Mobility Scale. In recent years, adjunctive technologies including electrical muscle stimulation, interactive video-games and passive cycle ergometry have also been utilised.

Delivery of early mobilisation is feasible, safe and effective in improving both short and long-term outcomes in critically ill patients even in the early stages of recovery whilst patients remain ventilated and receiving other forms of organ support. However, the optimum 'dose' of physical rehabilitation to deliver to patients whilst in the ICU remains undetermined. Early mobilisation reflects a clinically pragmatic approach to patient management, but there are few data to support the intensity, frequency and timing of interventions.

Furthermore, there is little known of the acute physiological response to undertaking this type of exercise in this patient population. Metabolic monitoring can provide information on the energy expenditure of patients. However, direct methods of data acquisition such as use of pulmonary artery catheters to measure whole-body oxygen consumption can be unreliable and their use in clinical practice has diminished in recent years. The non-invasive technique of indirect calorimetry (IC) has therefore emerged as a potential alternative that may be more practically applicable in the clinical setting. Indirect calorimetry measures total gas exchange, oxygen consumption and carbon dioxide production which can in turn determine energy expenditure. However the widespread clinical utility of the IC technique, can be offset by the number of clinical factors that may preclude its use across all patients e.g. those with cardiovascular or ventilator instability, those with open chest drainage or receiving renal haemofiltration.

Two studies to date have used IC to examine the response to physical rehabilitation activities performed by patients in the ICU. Collings et al conducted a randomised cross-over study in which 10 ICU patients completed either a passive chair transfer or an active sit-over-the-edge-of-the-bed (SOEOB) on one day, followed by the alternative activity on the consecutive day. The 'active' SOEOB activity elicited a significantly greater increase in oxygen consumption than the passive activity (90.69 ml/min (95% CI 44.04 to 137.34) vs 14.43 ml/min (95% CI -27.28 to 56.14), p = 0.007). Hickmann et al examined active or passive cycling in critically ill patients and healthy controls, demonstrating increased oxygen consumption during the active exercise compared to passive in patients with differing energy requirements compared to healthy individuals.

This limited existing evidence-base demonstrates the potential for use of IC to characterise physical rehabilitation in critically ill patients, but is restricted to particular types of activities and fails to capture sequential assessments of patients as their rehabilitation progresses through increasingly functional levels. Acknowledging the potential clinical limitations of applying the IC measurement technique to all critically ill patients, the aim of this study is to examine the feasibility of measuring energy expenditure of critically ill patients completing a range of physical rehabilitation activities (as characterised on the ICU Mobility Scale) performed sequentially during their ICU or ventilator weaning unit (Lane Fox Respiratory Unit, LFU) admission using indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Adult, ≥18years
* Receiving physical rehabilitation as part of routine physiotherapy management
* Invasively mechanically ventilated for ≥48hours
* Receiving invasive mechanical ventilation with stable settings

Exclusion Criteria:

* Endotracheal or tracheal leak >10%
* Burns
* Open chest drainage
* Inspired oxygen (FiO2) ≥0.6
* Extra-corporeal membrane oxygenation (ECMO)
* Pregnancy
* Cardiorespiratory instability requiring frequent adjustment of ventilator settings or FiO2, inotropic or sedative dosage, or positive end-expiratory pressure (PEEP) >10cmH2O
* Any neurological, orthopaedic or other factor contraindicating mobilisation
* Medical diagnosis mandating a specialist rehabilitation pathway e.g. amputee, acute neurological injury
* Palliative management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients undergoing physical rehabilitation in either the Intensive Care Units or the Lane Fox Unit at Guys and St Thomas' NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption during different physical rehabilitation activities. | Through Critical Care stay, an average of 1 per day
  Measurements of oxygen consumption during physical rehabilitation activities whilst on ICU
Carbon dioxide production during different physical rehabilitation activities. | Through Critical Care stay, an average of 1 per day
  Measurements of carbon dioxide production during physical rehabilitation activities whilst on ICU
Minute ventilation during different physical rehabilitation activities. | Through Critical Care stay, an average of 1 per day
  Measurements of minute ventilation during physical rehabilitation activities whilst on ICU

SECONDARY OUTCOMES:
Limitations of data acquisition using the indirect calorietry | Through Critical Care stay, an average of 9 days
  Measuring the quality of data acquired to identify technical issues, pragmatic factors, number of rehabilitation sessions by eligible patients and limiting factors to use of the indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Bronwen Connolly, Principal Investigator — Guys and St Thomas NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No